CLINICAL TRIAL: NCT06941207
Title: The Effect of Virtual Reality-Based Video and Benson Relaxation Exercise Applied to Palliative Care Providers on Sleep Quality, Fitness and General Well-Being
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, AHMET ŞİMŞEK, PhD student, Ataturk University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: ATAÜNİ-SBE-AS-01; ATATÜRK UNIVERSITY (Other: ATATÜRK UNIVERSITY SCIENTIFIC RESEARCH PROJECT UNIT)
Record Dates: First submitted 2025-04-10; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Palliative Care; Relaxation Therapy; Caregiver
Keywords: palliative care; benson relaxation exercise; virtual reality; sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- virtual reality video viewing group (Experimental): The first group in the experimental group, the virtual reality video group, caregivers, will be shown a total of 8 sessions of virtual reality-based videos (nature, forest walk and city tour, etc.) for an average of 30 minutes, twice a week for 4 weeks.
  Interventions: Behavioral: virtual reality video viewing group
- The group to which Benson relaxation exercise will be applied (Experimental): The second group in the experimental group, the caregivers, will have a total of 8 sessions of Benson relaxation exercises for 20-25 minutes, twice a week for 4 weeks.
  Interventions: Behavioral: benson relaxation exercise group
- control group (No Intervention): No intervention will be made to the caregivers in the control group.

INTERVENTIONS:
Behavioral: virtual reality video viewing group — The caregivers, the first group in the experimental group, will be shown a total of 8 sessions of virtual reality-based videos (nature, forest walks and city tours, etc.) for an average of 30 minutes, twice a week for 4 weeks.
  Arms: virtual reality video viewing group
Behavioral: benson relaxation exercise group — The second group in the experimental group, the caregivers, will have a total of 8 sessions of Benson relaxation exercises for 20-25 minutes, twice a week for 4 weeks.
  Arms: The group to which Benson relaxation exercise will be applied

SUMMARY:
The research will be conducted to evaluate the effects of Virtual Reality-Based Video and Benson Relaxation Exercise Applied to Palliative Care Providers on Sleep Quality, Fitness and General Well-Being. In the Palliative Care Center; The palliative patient group will be comprised of individuals aged 18 and over who provide care. The population of the research consists of 210 people. Individuals will be distributed to the virtual reality video experimental group (30), Benson relaxation exercise experimental group (30) and control (30) groups by simple randomization method. Personal Information Form, Sleep Quality Index, Subjective Wellness Scale and General Well-Being Scale will be used to collect research data. Personal information form, Sleep Quality Index, Subjective Well-Being Scale and General Well-Being Scale will be administered to the caregivers in both the experimental group and the control group by the researcher using face-to-face interview technique (pre-test).

The caregivers, the first group in the experimental group, will be shown a total of 8 sessions of virtual reality-based videos (nature, forest walks and city tours, etc.) for an average of 30 minutes, twice a week for 4 weeks.

The caregivers, who are the second group in the experimental group, will have a total of 8 sessions of Benson relaxation exercises for 20-25 minutes, twice a week for 4 weeks.

No intervention will be made to the caregivers in the control group. At the end of the sessions, Sleep Quality Index, Subjective Well-Being Scale and General Well-Being Scale (post-test) will be applied to the experimental and control groups.

The basic question it aims to answer is:

Do virtual reality-based video and BENSON relaxation exercises applied to palliative care givers affect sleep quality, vitality and general well-being?

DETAILED DESCRIPTION:
The word palliative originates from the Latin word "pallium", meaning "cover". What is intended to be achieved in palliative care is not to reduce the conditions that cause diseases or to prevent their development; but to reduce the problems that arise from diseases. The Role of Caregivers in Palliative Care; Their roles can be defined as individuals who are responsible for providing physical, economic, social and emotional support to the person receiving palliative care. The individual providing palliative care assumes the role of providing this communication and support during the medical, psychological and social support period. Providing care that does not require expertise; covers all needs such as meeting the nutritional needs of patients receiving palliative care, supporting their personal self-care needs, as well as providing special care to patients with tracheostomy, and feeding patients with PEG. Providing and performing palliative care is an action that is gained in a very different and multifaceted way for individuals providing palliative care. Although the job of providing care is stressful for palliative caregivers, in some ways, individuals providing care may perceive this action as a reward. As a result of this experience, the intimacy, love, personal communication skills and development of caregivers towards the patients they care for increase, and they can reach satisfaction during the care process. In addition to gaining positive experiences, palliative caregivers encounter many difficulties and challenges. In order to reduce or eliminate these difficulties, technological developments and classical methods should be used. Relaxation techniques, which are among the most important classical methods, are applied to various clinical problems such as childbirth, pain, insomnia, anxiety and aggression. Relaxation techniques reduce pulse, respiratory rate, blood pressure and oxygen consumption. Benson relaxation technique shows a protective mechanism against the fight or flight response that occurs in stress. When an individual is under stress, due to the increase in sympathetic nervous system activity; pulse, respiratory and metabolic rates increase, pupils dilate and vasoconstriction occurs. Stress hormones secreted for a long time and at high levels cause gastrointestinal system and cardiovascular system diseases, anxiety and sleep disorders. For this reason, Benson relaxation exercise tries to bring the body to the level it was before stress and prevent problems caused by stress hormones. In order to help protect and maintain health, which is one of the important issues of nursing, applications such as Benson relaxation exercise should be utilized. In addition, virtual reality applications in the field of health sciences are actively used in the protection stage of individuals before diseases occur, in the treatment process and rehabilitation stages, in the education, motivation and adaptation processes of students studying in these departments, employees providing health-related services, patients and individuals such as relatives and relatives who provide care to patients; and its area of use is expanding day by day. It has been revealed that with the increasing use of this and similar current technological aids in the field of health, it shortens the time spent on treatment by increasing the morale and motivation of patients and supports the information learned in student groups receiving education and training in health-related branches to be more effective and permanent. The importance of virtual reality-based educational models is as important and valuable as possible in the development of professional groups requiring manual skills and practice in students receiving education and training in medicine, health sciences and other branches, and in minimizing situations such as human-based medical errors. It is essential to use valuable and important virtual reality applications for caregivers to provide the necessary benefit. Palliative care takes a long time, the care burden is high, and caregivers experience difficulties in terms of physical, social and economic aspects. The majority of studies in the literature have been conducted on the determination of care burden and related factors. In a study conducted to determine the problems encountered by caregivers; 83.9% of the caregivers who participated in the study neglected themselves due to caregiving, 58.9% stated that their working life was negatively affected due to the illness and treatment process of the patient they cared for, 86.3% stated that their social life was negatively affected due to the caregiving process, 66.1% of the caregivers who participated in the study found that their health was negatively affected due to the caregiving process, 71% experienced sleep problems due to the illness and treatment process of their relative, 92.7% did not receive professional training on caregiving, and 54% needed psychosocial support due to the caregiving process. In order to solve the current situation, there are no studies that aim to reduce the negativities experienced by palliative caregivers. This study shows that virtual reality-based video application and Benson relaxation exercise applications will positively affect the sleep quality, vitality and general well-being of palliative caregivers, and this will both help caregivers maintain their health and provide better quality care to the patients they care for, thus reducing complications that may occur in patients, reducing the number of hospital admissions and producing positive economic results. In addition, the research is important in terms of contributing to the literature scientifically and providing resources for other research to be conducted on this subject.

Method The universe of the study will consist of individuals aged 18 and over who provide care to a palliative patient group admitted to Bilecik Bozüyük State Hospital Palliative Care Center. The universe of the study consists of 210 people. Individuals will be distributed to the virtual reality video experimental group (30), Benson relaxation exercise experimental group (30) and control (30) groups using a simple randomization method. Personal Information Form, Sleep Quality Index, Subjective Well-being Scale and General Well-being Scale will be used to collect the research data. Personal information form, Sleep Quality Index, Subjective Well-being Scale and General Well-being Scale will be applied to the caregivers in both the experimental and control groups by the researcher using face-to-face interview technique (pre-test).

The caregivers in the first group in the experimental group will be shown a total of 8 virtual reality-based videos (nature, forest walk and city tour etc.) for an average of 30 minutes, twice a week for 4 weeks.

The second group in the experimental group, the caregivers, will have 8 sessions of Benson relaxation exercises, 20-25 minutes twice a week for 4 weeks.

No intervention will be made to the caregivers in the control group.

At the end of the sessions, the Sleep Quality Index, Subjective Vitality Scale and General Well-Being Scale (post-test) will be applied to the experimental and control groups.

Targets to be achieved Virtual reality-based video is an easily applicable, simple application, and it aims to maintain the health of palliative caregivers and increase their quality of life by making positive contributions to palliative caregivers, by positively affecting their sleep quality, vitality and general well-being.

Benson relaxation exercise application is an easily applicable, free and simple application, and it aims to provide positive contributions to palliative caregivers, by positively affecting their sleep quality, vitality and general well-being, both to maintain the health of palliative caregivers and to provide more effective care to the patient group they provide care for, thus reducing repeated applications to health institutions and making positive contributions in economic terms.

Since neither application has side effects, it is aimed to be adopted and widespread as a new non-pharmacological method by palliative caregivers and nurses.

The effect of virtual reality-based video and Benson relaxation exercise applications on sleep quality, vitality and general well-being for palliative caregivers shows that the project has original value, and it is aimed that the project results will contribute to national and international literature. It is anticipated that virtual reality-based video and Benson relaxation exercise applications applied to palliative caregivers will have a positive effect on sleep quality, vitality and general well-being.

ELIGIBILITY:
Inclusion Criteria:

1. Being literate,
2. Being over the age of 18,
3. Having sufficient communication skills to answer oral and written questions and follow instructions,
4. Being a palliative care provider for at least 6 months
5. Does not have visual/verbal/auditory communication difficulties that would prevent understanding the information presented and expressing the answers correctly,
6. Being a caregiver who can communicate in Turkish
7. Not having severe vision problems

Exclusion Criteria:

1. Sleep Quality Index score of 4 or less
2. Being over 65 years old
3. Palliative care providers who leave the study voluntarily
4. Presence of chronic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 1 month
  PSQI, developed by Buysse et al. (1989) and validated and reliable in Turkish by Ağargün (1996), is a self-report-based assessment tool that provides information about sleep quality and the type and severity of sleep disorders in the last month.
subjective fitness scale | 1 month
  Subjective Wellness Scale (SWS) is a scale developed by Ryan and Frederick in 1997. The adaptation of the scale to Turkish and its validity and reliability studies were conducted by Uysal et al. (2014). ESS is a self-report measuring tool consisting of 7 items and on a 7-point Likert scale (1 strongly disagree - 7 strongly agree).
General Well-Being Scale Short Form | 1 month
  The General Well-Being Scale, developed by Longo et al. (2018) and adapted into Turkish by Odacı et al. (2021), consists of 14 items that aim to measure the person's affect and satisfaction level with his life. Within the scope of the validity studies of the scale, confirmatory factor analysis, correlational analysis and independent samples t test were performed. According to the results of the factor analysis, it was confirmed that the scale had a single-factor structure. As a result of the criterion-related validity analysis, a significant positive relationship was detected between the participants' general well-being levels and positive affect, their life satisfaction and their needs satisfaction; A significant negative relationship was detected between negative emotions and negative emotions.